CLINICAL TRIAL: NCT02436031
Title: The Effect of Desipramine on Upper Airway Collapsibility and Genioglossus Muscle Activity During Sleep in Patients With Obstructive Sleep Apnea - Study B
Brief Title: Effect of Desipramine on Upper Airway Collapsibility and Genioglossus Muscle Activity in Patients With Obstructive Sleep Apnea - Study B
Acronym: DESOSA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, David Andrew Wellman, Assistant Professor of Medicine, Harvard Medical School | Director, Sleep Disordered Breathing Lab, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BWH-2014P001033B
Record Dates: First submitted 2015-05-01; First posted 2015-05-06 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Desipramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desipramine First, Placebo Second (Active Comparator): Desipramine 200 mg administered 2 hours before normal sleep time on first study night, then a 1-week non-treatment period, then placebo-matching desipramine administered 2 hours before normal sleep time on second study night.
  Interventions: Drug: Desipramine; Drug: Placebo
- Placebo First, Desipramine Second (Experimental): Placebo-matching desipramine administered 2 hours before normal sleep time on first study night, then a 1-week non-treatment period, then desipramine administered 2 hours before normal sleep time on second study night.
  Interventions: Drug: Desipramine; Drug: Placebo

INTERVENTIONS:
Drug: Desipramine — 200 mg administered 2 hours before normal sleep time
  Other Names: Norpramine
Drug: Placebo — Placebo-matching desipramine administered 2 hours before normal sleep time

SUMMARY:
Obstructive sleep apnea (OSA) is common and has major health implications but treatment options are limited. OSA patients show a marked reduction in upper airway (UA) dilator muscle activity at sleep onset and this phenomenon leads to increased collapsibility of UA compared to normal participants. Until recently, the search for medicines to activate pharyngeal muscles in sleeping humans has been discouraging. However, exciting new animal research has shown that drugs with noradrenergic and antimuscarinic effects can restore pharyngeal muscle activity to waking levels. In this protocol the investigators will test the effect of desipramine (a tricyclic antidepressant with strong noradrenergic and antimuscarinic effects) on upper airway collapsibility and genioglossus muscle activity (EMG GG) during sleep in OSA patients.

DETAILED DESCRIPTION:
Two overnight sleep studies, a placebo night and a drug night, will be performed approximately one week apart in random order. The placebo or drug will be administered 2 hours before lights out. At least 15 minutes of quiet wakefulness will be recorded to quantify the participant's EMG GG activity while awake and at sleep onset (alpha-theta transition at the electroencephalogram).

During the second part of the night, the participants will be connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which can provide a wide range of pressures between 20 and -20 cmH2O in order to modify upper airway pressure and measure pharyngeal critical collapsing pressure (Pcrit), ventilation at 0 cmH2O when UA muscle are passive and active as well as change in EMG GG as a function of epiglottic pressure (muscle responsiveness).

Apnea-hypopnea index (AHI) will be calculated in each night from the part of the study off CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed OSA (moderate-to-severe; apnea hypopnea index >15 events/hr)

Exclusion Criteria:

* Cardiovascular disease other than well controlled hypertension
* Depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Wellman, MD PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Sleep Disorders Research Program Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: First Study Night
Arm/Group | Desipramine First, Placebo Second | Placebo First, Desipramine Second
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Second Study Night
Arm/Group | Desipramine First, Placebo Second | Placebo First, Desipramine Second
Started | 7 (1 participant did not tolerate the study setup so did not participate in the second study night) | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Analyzed Participants: All participants who were randomized, completed both study nights, and were included in the analysis. 1 participant was excluded due to insufficient sleep time.
Arm/Group | All Analyzed Participants
Number analyzed (Participants) | 14
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [49 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Pharyngeal Critical Collapsing Pressure (Pcrit) as a Measure of Upper Airway Collapsibility
Description: Participants were connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which provided a wide range of pressures between 20 and -20 cm H2O in order to modify upper airway pressure. Following a baseline recording period of 5 minutes, the CPAP level was reduced to varying suboptimal pressures. Change in Pcrit was used to determine the collapsibility of the upper airway under both passive and active conditions, and is expressed as Passive Pcrit: ventilation at a nasal pressure of 0 cm H2O when pharyngeal muscles are passive; Active Pcrit: ventilation at a nasal pressure of 0 cm H2O when pharyngeal muscles are active. Improved=more negative Pcrit.
Time Frame: 1 night
Population: All participants who were randomized, completed both study nights, and were included in the analysis. 1 participant was excluded due to insufficient sleep time.
Measure: Median (Inter-Quartile Range); unit: cm H2O
Groups:
- Desipramine: Desipramine 200 mg administered 2 hours before normal sleep time on the first study night or second study night.
- Placebo: Placebo-matching desipramine administered 2 hours before normal sleep time on the first study night or second study night.
Arm/Group | Desipramine | Placebo
Number analyzed (Participants) | 14 | 14
cm H2O
  Active Pcrit | -5.2 [-7 to -2.8] | -1.9 [-3.3 to -0.7]
  Passive Pcrit | -2.2 [-3.2 to 0.2] | -0.7 [-1.7 to -0.4]
Statistical Analysis 1: Comparison: Desipramine vs Placebo; Active Pcrit; Test type: Other; p = 0.049, Wilcoxon Matched-Pairs Signed-Rank Test
Statistical Analysis 2: Comparison: Desipramine vs Placebo; Passive Pcrit; Test type: Other; p = 0.135, Wilcoxon Matched-Pairs Signed-Rank Test

2. Secondary Outcome: Genioglossus Muscle Responsiveness to Progressively Greater Epiglottic Pressure Swings
Description: Electromyography (EMG) was used to analyze genioglossus (GG) [EMG GG] muscle activity. EMG GG activity was recorded via standard needle electrodes inserted into the genioglossus muscle (tongue). Activity of EMG GG was measured during wakefulness and sleep as % of maximum activation obtained pushing the tongue against closed teeth during wakefulness (GG%max). Participants were connected to a modified continuous positive airway pressure (CPAP) machine (Pcrit3000, Respironics) which provided a wide range of pressures between 20 and -20 cm H2O in order to modify upper airway pressure and measure change in EMG GG as a function of epiglottic pressure (muscle responsiveness) (%max/cmH2O).
Time Frame: 1 night
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: %max/cmH2O
Arm/Group | Desipramine | Placebo
Number analyzed (Participants) | 14 | 14
%max/cmH2O | -0.24 [-0.5 to -0.2] | -0.25 [-0.4 to -0.1]

3. Secondary Outcome: Number of Apnoea-Hypopnea Index (AHI) Events During Non-Random Eye Movement (NREM) Sleep
Description: The AHI is the number of apneas (pauses in breathing) or hypopneas (shallow breathing) recorded during the study per hour of sleep. Data for the calculation of the AHI was collected while the participant was in NREM sleep in the supine position and off CPAP (breathing spontaneously).
Time Frame: 1 night
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: events per hour
Arm/Group | Desipramine | Placebo
Number analyzed (Participants) | 13 | 13
events per hour | 34.3 [14.7 to 62] | 42.0 [20.5 to 53.3]

ADVERSE EVENTS:
Description: All randomized participants who received at least one dose of desipramine or placebo.
Arm/Group | Desipramine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 1/16 | 0/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Desipramine (N=16) | Placebo (N=15)
Dizziness (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes